CLINICAL TRIAL: NCT05135143
Title: Role of Antioxidants in the Reduction of Oxidative Stress in Infertile Patients
Acronym: OAT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Tetova (Other)
Collaborators: University of Tetova, Faculty of Medical Sciences (Unknown)
Responsible Party: Principal Investigator, Vegim Zhaku, Medical Doctor and Teaching assistant, University of Tetova
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 22-63/3
Record Dates: First submitted 2021-10-25; First posted 2021-11-26 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Infertility; Oligoasthenozoospermia; Male
Keywords: antioxidant; oxidative stress; sperm parameters; Malonedialdehyde; total antioxidant capacity
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Double blind randomized
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Infertility male patients (Active Comparator): Infertile male patients will receive the antioxidant formula for more than 172 days. Divided in two groups. One will take the active substance, to the other group placebo treatment will be given.
  Interventions: Combination Product: Antioxidant formula
- Control group (Placebo Comparator): Placebo treatment and control and comparative variables will be measured.
  Interventions: Combination Product: Antioxidant formula

INTERVENTIONS:
Combination Product: Antioxidant formula — Administration of antioxidant formula 3 times a day and once daily.

SUMMARY:
Numerous studies verify that the majority of cases of male infertility belong to the group diagnosed with oligoasthenoteratozoospermia (OAT), which means a decrease in the number of sperm in the ejaculate to 15 million / ml, reduced sperm motility of the spermatozoa and morphological disorders of the neck or tail of the sperm.

Genuine scientific studies can not pinpoint the cause of these changes, however, recent advances in science shed light on this issue by confirming the reason, which is as a result of the action of free radicals - oxidative stress.

DETAILED DESCRIPTION:
The enlightenment project in the field of male infertility in North Macedonia will include a wide team of: students, general practitioners, assistants, professors of pre-clinical subjects, professors and specialists in the field of gynecology, urology and andrologists. The involvement of such a large number of professionals once again verifies the seriousness and determination that this scientific project has.

Investigators hope to contribute generously to:

1. Identifying new cases and taking measures early, in order to overcome fertilization problems;
2. For the first time in North Macedonia there will be a more accurate picture of the prevalence of male infertility;
3. Expanding current scientific knowledge about the role of oxidative stress, its laboratory evaluation, and the impact of antioxidant supplements;
4. Standardization of doses and type of antioxidant supplements that will be used during the realization of this dissertation and evaluation of their clinical effect in men with OAT;
5. After the implementation of antioxidant therapy, investigators expect that the results of live births and spontaneous pregnancies will increase, while the number of miscarriages will decrease;
6. Acquisition of knowledge on laboratory and clinical evaluation techniques of infertile men, which would later lead to the establishment of an andrological laboratory. Investigators anticipate this laboratory to function within the Faculty of Medical Sciences, where all procedures will be performed, from diagnosis to the operation of assisted reproduction techniques (TRA). This, in addition to the material benefit for the benefit of the University of Tetova, also has a benefit in terms of staff, which will be professionalized and trained during the realization of this dissertation.

ELIGIBILITY:
Inclusion Criteria:

* age, 19-45 years;
* infertility, 2 years;
* regular sexual intercourse with a fertile female.
* The female partner was defined as being fertile if she had undergone a negative infertility workup (biphasic basal body temperature, P evaluation in luteal phase, ultrasound ovary and uterus evaluation, and hysterosalpingogram to study tubal patency)

Exclusion Criteria:

* use of antioxidant agents or vitamins within 8 weeks prior to inclusion in the study,
* a history of excessive consumption of alcohol 40 days prior to the start of the trial,
* patients that showed lower than 5% motility and less than 1 × 106/ml sperm concentration, - patients with any acute or chronic disease or
* who are undergoing some kind of treatment with any class of drugs and
* subjects with known hypersensitivity to ingredients in the antioxidant formula.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Because investigators have to measure sperm parameters
Enrollment: 211 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Sperm parameters | 6 months
  Concentration (10x6 ml)
Sperm parameters | 6 months
  Morphology (percentage)
Sperm parameters | 6 months
  Motility (percentage)

SECONDARY OUTCOMES:
oxidative stress parameters | 6 months
  MDA (mg/ml)
oxidative stress parameters | 6 months
  Caspase 3 (IU/ml)
oxidative stress parameters | 6 months
  TAC (IU/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Vegim Zhaku, MD, PhDc, Principal Investigator — University of Tetova; Sheqibe Beadini, PhD, Study Chair — University of Tetova; Nexhbedin Beadini, PhD, Study Chair — Univeristy of Tetova
Locations (1):
- Univeristy of Tetova, Tetovo, North Macedonia

IPD SHARING:
Plan to Share IPD: Undecided
Sperm parameters before and after treatment. OS parameters before and after treatment.

REFERENCES:
- [Background] Vegim Zhaku, Ashok Agarwal, Sheqibe Beadini, Ralf Henkel, Renata Finelli, Nexhbedin Beadini and Sava Micic (June 8th 2021). Male Infertility, Oxidative Stress and Antioxidants, Vitamin E in Health and Disease - Interactions, Diseases and Health Aspects, Pınar Erkekoglu and Júlia Scherer Santos, IntechOpen, DOI: 10.5772/intechopen.98204. Available from: https://www.intechopen.com/chapters/77097
- [Background] ] Zhaku V, Beadini Sh, Beadini N, Xhaferi V, Golaboska J. The role of semen analysis in the expression of male infertility in southwestern part of North Macedonia (Experiences from 7 municipalities). UNIVERSI-International Journal of Education Science Technology Innovation Health and Enviroment. 2019;5(2):96-104.
- [Background] Zhaku V, Beadini Sh, Beadini N, Murtezani B. Combination of Maca, Korean ginseng extract and antioxidant therapy for male with oligoasthenozoospermia: case study. Journal of Hygienic Engineering and Design. 2019; 26(1):28-35.
- [Background] Zhaku V, Beadini Sh, Beadini N, Xhaferi V. Role of antioxidants in the diminution of oxidative stress and amelioration of semen parameters in idiopathic male infertility. Acta Medica Balkanica. 2020; 5(9-10):69-80.
- [Background] Zhaku V, Beadini Sh, Beadini N, Xhaferi V, Milenkovic T. Oral antioxidants improve sperm motility, sperm concentration and reduce oxidative stress in males with oligo-asthenozoospermia. In: 22nd European Congress of Endocrinology; 5-9 September 2020; Prague, Czech Republic: Endocrine Abstracts (2020) 70 EP581. DOI:10.1530/ endoabs.70.EP581
- See also: Male infertility, Oxidative Stress and Antioxidants — https://www.intechopen.com/chapters/77097
- See also: ROLE OF ANTIOXIDANTS IN THE DIMINUTION OF OXIDATIVE STRESS AND AMELIORATION OF SEMEN PARAMETERS IN IDIOPATHIC MALE INFERTILITY — https://eprints.unite.edu.mk/561/
- See also: COMBINATION OF MACA, KOREAN GINSENG EXTRACT AND ANTIOXIDANT THERAPY FOR MALE WITH OLIGOASTHENOZOOSPERMIA: CASE STUDY — https://keypublishing.org/jhed/jhed-volumes/jhed-volume-26-fqs-3-vegim-zhaku-sheqibe-beadini-nexhbedin-beadini-besir-murtezan-2019-combination-of-maca-korean-ginseng-extract-and-antioxidant-therapy-for-male-with-oligoasthenozoos/
- See also: Oral antioxidants improve sperm motility, sperm concentration and reduce oxidative stress in males with oligoasthenozoospermia — https://www.endocrine-abstracts.org/ea/0070/ea0070ep581